CLINICAL TRIAL: NCT01810796
Title: Pathophysiology and Prevention of Perioperative Myocardial Injury: A Prospective Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Giora Landesberg, Associate Profesor, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HRanTrop
Record Dates: First submitted 2013-03-12; First posted 2013-03-14 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Coronary Artery Disease,
MeSH Terms: conditions — Coronary Artery Disease | interventions — Ranolazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ranolazine treatment (Experimental): Ranolazine 500-1000mg bid
  Interventions: Drug: Ranolazine
- Placebo (Placebo Comparator): Placebo

INTERVENTIONS:
Drug: Ranolazine — Ranolazine versus placebo
  Other Names: Ranexa
  Arms: Ranolazine treatment

SUMMARY:
Working hypothesis and aims: 1) To explore the pathophysiology of postoperative troponin elevations and 2) whether ranolazine, a new anti-ischemic drug that has no effect on blood pressure or heart rate, prevents postoperative myocardial injury.

DETAILED DESCRIPTION:
High-risk patients undergoing non cardiac surgery will be randomized to receive either Ranolazine or placebo perioperatively and troponin will be measured on the first 3 days after surgery.

ELIGIBILITY:
Inclusion Criteria:

- All patients age 18 and above, undergoing major surgery that require at least 24 hours (overnight) stay in the post anesthesia care unit (PACU) or intensive care unit (ICU), and who either have known history of CAD or at least 3 of the following Revised Cardiac Risk Index (RCRI) criteria29F17: 1) high-risk type of surgery, 2) history of ischemic heart disease, 3) history of congestive heart failure, 4) history of cerebrovascular disease, 5) diabetes mellitus, 6) renal failure (creatinine > 2mg/ml).

Exclusion Criteria:

* Pregnancy, LV ejection fraction ≤35%, patients with severe valvular disease, patients with poor echocardiographic images, patients who cannot swallow the pill after surgery, refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2013-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Postoperative troponin | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Giora Landesberg, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah - Hebrew University Medical Center, Jerusalem, Israel